CLINICAL TRIAL: NCT01622660
Title: Phase II Study of Gemcitabine and Pazopanib in Chemotherapy Naïve Patients With Advanced/Metastatic Urothelial Carcinoma Ineligible for Cisplatin-based Chemotherapy
Brief Title: Gemcitabine and Pazopanib in Chemotherapy Naïve Patients With Advanced/Metastatic Urothelial Carcinoma Ineligible for Cisplatin-based Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety reasons
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-191
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-05

CONDITIONS: Bladder Cancer
Keywords: URETER; URINARY BLADDER; renal pelvis; GEMCITABINE; GW786034 (PAZOPANIB); 11-191
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; pazopanib

ARMS (1):
- Gemcitabine and Pazopanib (Experimental): This is a phase II trial of gemcitabine and pazopanib in previously untreated patients with advanced/metastatic urothelial carcinoma (UC) who are ineligible for cisplatin-based chemotherapy.
  Interventions: Drug: Gemcitabine; Drug: Pazopanib

INTERVENTIONS:
Drug: Gemcitabine — Patients will receive gemcitabine 1200 mg/m2 intravenously on day 1 and day 8 and. Patients will receive 6 cycles of combination therapy (gemcitabine and pazopanib) unless disease progression or unacceptable toxicity occurs. Patients that achieve stable disease, a partial response, or a complete response after completion of 6 cycles, and who are not candidates for consolidation surgery, will be eligible to continue pazopanib monotherapy at the same dose and schedule until disease progression for a maximum of 18 additional cycles.
Drug: Pazopanib — pazopanib 800 mg orally daily day 1 through day 21 (1 cycle = 21 days) Patients will receive 6 cycles of combination therapy (gemcitabine and pazopanib) unless disease progression or unacceptable toxicity occurs. Patients that achieve stable disease, a partial response, or a complete response after completion of 6 cycles, and who are not candidates for consolidation surgery, will be eligible to continue pazopanib monotherapy at the same dose and schedule until disease progression for a maximum of 18 additional cycles.

SUMMARY:
Gemcitabine and Cisplatin are standard chemotherapy drugs used to treat advanced urothelial cancer. There is no standard chemotherapy for patients who cannot receive Cisplatin. However, most patients are treated with the chemotherapy drugs Gemcitabine and Carboplatin.

In this study, the researchers hope to learn what effects, good and/or bad, the combination of Gemcitabine and Pazopanib has on urothelial cancer. Gemcitabine is given intravenously (through the veins) and works by killing rapidly dividing cells in the body, including cancer cells. Pazopanib is an oral chemotherapy and works by decreasing the blood supply to tumors which limits the tumor's source of oxygen and nutrients.

The combination of Gemcitabine and Pazopanib is being tested in research studies such as this one. As of August 2011, more than 18 patients with various types of cancer have received treatment with Gemcitabine and Pazopanib. The main goal of this clinical research study is to learn if the study drugs Gemcitabine and Pazopanib can shrink or slow the growth of urothelial cancer. The safety of this drug will also be studied. The physical state, changes in the size of the tumor, and laboratory findings will help us decide if the combination of Gemcitabine and Pazopanib is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis by MSKCC pathology review
* Measurable disease as determined by RECIST v1.1 on initial pretreatment staging CT scan of the chest, abdomen, and pelvis (or MRI if clinically appropriate). (Note: A chest x-ray may be performed as an alternative to a CT scan of the chest.)
* Ineligible for cisplatin based on one or more of the following:

  * Calculated creatinine clearance of < 60 mL/min (but ≥ 30 mL/min)
  * Karnofsky Performance Status (KPS) 60-70% (ECOG PS 2)
  * Grade 2 ≥ hearing loss
  * Grade 2 ≥ peripheral neuropathy
* Karnofsky Performance Status ≥ 60%
* 10 unstained slides or paraffin embedded tissue block obtained from pretreatment tumor specimens for immunohistochemistry. (Note: One paraffin block or 10 freshly-prepared unstained slides from the most representative single paraffin embedded tumor tissue block should be submitted. Slides from the primary tumor are preferred. If both the primary and metastatic tumor blocks are available, 10 slides from each of the sites should be submitted. If tissue from the primary tumor is not available, a paraffin block or unstained slides from a metastatic site are acceptable. Fine needle aspirates (FNAs) have insufficient tumor tissue and are not permitted.)
* Adequate organ system function as defined:

  * Absolute neutrophil count (ANC) ≥1.5 X 109/L
  * Hemoglobin ≥9 g/dL (5.6 mmol/L) (Note: Subjects may not have had a transfusion within 7 days of screening assessment.)
  * Platelets ≥100 X 109/L
  * Prothrombin time (PT) or international normalized ratio (INR) ≤1.2 X ULN (Note: Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.)
  * Activated partial thromboplastin time (aPTT) ≤1.2 X ULN
  * Total bilirubin ≤1.5 X ULN
  * Alanine amino transferase (ALT) and Aspartate aminotransferase (AST)

    ≤2.5 X ULN (Note: Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted.)
  * Calculated creatinine clearance (ClCR) ≥30 mL/min using the CKD-EPI equation: eGFR = 141 x min(Scr/k, 1)a x max(Scr/k, 1)-1.209 x 0.993 Age x 1.018 [if female] x 1.159 [if black] Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is - 0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1
  * Urine Protein to Creatinine Ratio (UPC)d <1 (Note: If UPC ≥1, then a 24- hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1 g to be eligible.)

Exclusion Criteria:

* Prior treatment with systemic chemotherapy (prior intravesical therapy is permitted)
* Prior malignancy (Note: Subjects who have had another malignancy and have been disease-free for 5 years subjects with a history of completely resected non-melanomatous skin carcinoma, subjects with successfully treated in situ carcinoma, or subjects who have had adenocarcinoma of the prostate that has been definitively treated with a post-treatment PSA that is non-detectable are eligible.)
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:
  * Malabsorption syndrome
  * Major resection of the stomach or small bowel
* Active liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
* Presence of uncontrolled infection Corrected QT interval (QTc) > 480 msecs using Bazett's formula

  o If QTc interval is > 480 msecs, then 2 additional ECGs should be obtained over a brief period of time (e.g., within approximately 15-20 minutes) to confirm the abnormality. The average QTc interval will be determined from the 3 ECG tracings by manual evaluation and will be used to determine if the subject will be excluded from the study. If the average QTc interval is >480 msec, then the subject is not eligible to participate in the study Previous history of QTc prolongation as a result of other medication that required discontinuation of that medication
* Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age
* Use of any concomitant medication (during treatment with pazopanib or within 14 days of starting treatment) that are high risk for QTc prolongation or may induce Torsades de Pointes.
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction Unstable angina
  * Coronary artery bypass graft surgery
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg] (Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. At least 24 hours after initiation or adjustment of antihypertensive medication (s), BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP / DBP values from each BP assessment must be <140/90 mmHg in order for a subject to be eligible for the study.)
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. (Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.)
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Evidence of active bleeding or bleeding diathesis. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications listed in (Concomitant Therapy) for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
* Treatment with any of the following anti-cancer therapies:

  * Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR
  * Immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity
* Women who are pregnant or breast feeding (Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.)
* Adults of child-bearing potential not employing an effective method of birth control for two weeks prior to study start and 21 days after the last dose. All women of child-bearing potential must have a negative serum pregnancy test. Women of child-bearing potential are defined as sexually mature women who have not undergone a hysterectomy, bilateral oophorectomy (ovariectomy), or bilateral tubal ligation OR have not experienced total cessation of menses for ≥ 1 year and are older than 45 years in age, In questionable cases, the patient must have a follicle stimulating hormone (FSH) value >40 mIU/mL and an estradiol value < 40pg/mL (<140 pmol/L). Effective methods of birth control are defined in section 9.9 (Contraception Requirements).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Bajorin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 06/14/2012 Protocol Closed to Accrual 02/05/2014 Primary Completion Date 02/03/2016 Recruitment Location is the medical clinic
Groups:
- Gemcitabine and Pazopanib: Chemotherapy naïve participants with advanced/metastatic urothelial carcinoma ineligible for Cisplatin-based chemotherapy
Period: Overall Study
Arm/Group | Gemcitabine and Pazopanib
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine and Pazopanib: This is a phase II trial of gemcitabine and pazopanib in previously untreated patients with advanced/metastatic urothelial carcinoma (UC) who are ineligible for cisplatin-based chemotherapy.
  Gemcitabine and Pazopanib: Patients will receive gemcitabine 1200 mg/m2 intravenously on day 1 and day 8 and pazopanib 800 mg orally daily day 1 through day 21 (1 cycle = 21 days). Patients will receive 6 cycles of combination therapy (gemcitabine and pazopanib) unless disease progression or unacceptable toxicity occurs. Patients that achieve stable disease, a partial response, or a complete response after completion of 6 cycles, and who are not candidates for consolidation surgery, will be eligible to continue pazopanib monotherapy at the same dose and schedule until disease progression for a maximum of 18 additional cycles.
Arm/Group | Gemcitabine and Pazopanib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 70.5 [60 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival will be calculated from the start of treatment until progressive disease or death. Patients who die before documented progression will be considered failures at their time of death. If the patient did not progress or die, the patient will be censored on the date of last follow-up. Response and progression will be evaluated in this study using the international criteria by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 Measurable lesions: lesions that can be accurately measured in at least one dimension with longest diameter ≥ 10 mm by clinical exam or with spiral CT scan or MRI (no less than double the slice thickness and a minimum of 10mm). Malignant lymph nodes must be 15 mm in the short axis when assessed by spiral CT scan to be considered measurable. Non-measurable lesions: all other lesions (or sites of disease) including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm u
Time Frame: 2 years
Measure: Number; unit: days
Arm/Group | Gemcitabine and Pazopanib
Number analyzed (Participants) | 1
days | 184

ADVERSE EVENTS:
Time Frame: 0.8 months to 6.3 months
Description: Adverse event data were collected for the duration of treatment. For Patient 001 this was 0.8 months. For Patient 002 this was 6.3 months.
Arm/Group | Gemcitabine and Pazopanib
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Pazopanib (N=2)
Elevated ALT with concomitant elevation in Bilirubin (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine and Pazopanib (N=2)
Elevated ALT (Hepatobiliary disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Elevated AST (Hepatobiliary disorders) | 1
Blood Bilrubin Increased (Hepatobiliary disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Gastroesophageal reflux disorder (Gastrointestinal disorders) | 1
Gastrointestinal disorders, other (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
INR increased (Investigations) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Leukopenia (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes